CLINICAL TRIAL: NCT02435654
Title: Effects of 5-HTR2A, DRD2,and COMT Genes Polymorphisms and Drug Plasma Concentration on Antipsychotic Response to Olanzapine in Treatment of Early-onset Schizophrenia
Brief Title: 5-HTR2A, DRD2,and COMT Genes Polymorphisms and Olanzapine Plasma Concentration in Treatment of Early-onset Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kunming Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Kang Chuanyuan, chief physician, Kunming Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81460218
Record Dates: First submitted 2015-04-28; First posted 2015-05-06 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2019-09

CONDITIONS: Early-onset Schizophrenia
Keywords: Genes Polymorphisms; Plasma Concentration
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): All EOS patients will receive olanzapine treatment with flexible dose(2.5 to 20 mg/day)according to standard body weight,olanzapine will be initiated at 2.5 or 5 mg/day and the dose could be increased by 2.5 or 5 mg/day dose increments at the investigator's discretion.A effective dose would be titrated in two weeks with no tolerability or safety issues are apparent,the investigator could decrease the dose at any time and in any number of dose decrements if patients experienced an adverse event.
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — olanzapine will be initiated at 2.5 or 5 mg/day according to patient's weight, and the dose could be increased by 2.5 or 5 mg every 4-7days at the investigator's discretion.A effective dose would be titrated in two weeks with no tolerability or safety issues are apparent,
  Other Names: Zyprexa

SUMMARY:
In this study,investigators will recruit 100 DSM-Ⅴdefined EOS Han patients, older than 7 years old and onset of illness before 17 years old, and all EOS patients will receive a 8-week systematic olanzepine titration treatment and a battery of assessments of treatment effect and safety. Blood olanzepine plasma concentration will be tested regularly and genotyping of 8 polymorphisms of 5-HTR2A, DRD2 and COMT genes will be conducted by Polymerase Chain Reaction （PCR）, Restriction Fragment Length Polymorphism (RFLP) and TaqMan probes genotyping technology. The aim of the study is to explore the predictive factors on olanzepine treatment response in EOS, which can guide the individualized treatment and improve the cure rate of EOS in clinical setting.

DETAILED DESCRIPTION:
Early-onset schizophrenia (EOS) is the World Health Organization ranked psychosis as the third most disabling condition worldwide in youth, and may lead to obvious social dysfunction and interfere seriously with neurodevelopmental processes in a young person, which in turn has the potential to irreversibly alter the trajectory of his or her life. To improve the outcome of the patients of EOS, elaborate and individualized therapeutic regimen is urgently needed. The functional gene polymorphisms and drug (antipsychotics) plasma concentration can both influence the drug response, but few studies explore the contributions of genetic heterogeneity, drug plasma concentration and clinical features of patients to drug response together and interactions of above factors in EOS patients. In this study investigators will recruit 100 DSM-Ⅴdefined EOS Han patients, older than 7 years old and onset of illness before 17 years old, and all EOS patients will receive a 8-week systematic olanzepine titration treatment and a battery of assessments of treatment effect and safety. Blood olanzepine plasma concentration will be tested regularly and genotyping of 8 polymorphisms of 5-HTR2A, DRD2 and COMT genes will be conducted by Polymerase Chain Reaction （PCR）, Restriction Fragment Length Polymorphism (RFLP) and TaqMan probes genotyping technology. The aim of the study is to explore the predictive factors on olanzepine treatment response in EOS, which can guide the individualized treatment and improve the cure rate of EOS in clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* above 7 years old,
* age of onset ≤17 years old,
* Han or other nationality, male or female,
* in line with the diagnostic DSM-V criteria for schizophrenia, and
* negative and positive symptom scale (Positive and Negative Syndrome Scale, PANSS) score ≥70 points;
* patients are in the condition of first-episode, or relapse.

Exclusion Criteria:

* IQ <70,
* current or previous history of traumatic brain injury,
* psychoactive substance use,
* personality disorders,
* obvious abnormalities on physical and laboratory examination,
* previous allergy or olanzapine had significant adverse reactions.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
multiple regression equation of 5-HTR2A、DRD2 and COMT Genes Polymorphisms and Olanzapine Plasma Concentration and clinical features | 12 weeks

SECONDARY OUTCOMES:
change in score of PANSS | baseline and 12 weeks
plateau concentration of olanzapine | 2 or 3,12 weeks
change in Serum prolactin levels | 12 weeks
Prevalence associated with age、gender and onset form | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu xiufeng, Principal Investigator — Psychiatry Department ,First Affiliated Hospital Of Kunming Medical University
Locations (1):
- Psychiatry Department,First Affiliated Hospial Of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No